CLINICAL TRIAL: NCT00207779
Title: Prevention of Catheter-Related Bloodstream Infection in Patients With Haemato-Oncological Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre National de Greffe de Moelle Osseuse (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E02
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Infection
Keywords: central venous catheter; catheter related bloodstream infection; heparin
MeSH Terms: conditions — Infections

INTERVENTIONS:
Device: heparin impregnated central venous catheters

SUMMARY:
We, the researchers at Centre National de Greffe de Moelle Osseuse, have shown in a randomised study (in press), that a low dose of unfractionated heparin (100 IU/kg/daily) was safe and effective to prevent catheter-related bloodstream infection in patients with haemato-oncological disease.

The aim of this prospective randomised controlled trial is to compare the incidence of catheter-related bloodstream infection in 2 groups of patients with haemato-oncological disease:

* Group A: heparin impregnated catheters
* Group B: low-dose unfractionated heparin (100 IU/kg/daily)

DETAILED DESCRIPTION:
Studies have shown that catheter-related infection may be due to fibrin deposition associated with catheters. Interventions designed to decrease fibrin deposition and thrombus formation have the potential to reduce catheter-related infections. Seven randomised studies have been performed to assess the safety and efficacy of heparin (either as an infusion or bonded to central venous catheter) on central venous catheter-related bloodstream infections. Although a meta-analysis of 4 studies looking at heparin either as an infusion or bonded to central venous catheter showed a strong trend for a reduction in catheter-related bloodstream infection with the use of heparin, these studies used variable definitions of catheter-related infections.

We have shown in a randomised study (in press), that low dose of unfractionated heparin (100 IU/kg/daily) was safe and effective to prevent catheter-related bloodstream infection in patients with haemato-oncological disease. The aim of this prospective randomised controlled trial is to compare the incidence of catheter-related bloodstream infection in 2 groups of patients with haemato-oncological disease:

* Group A: heparin impregnated catheters
* Group B: low-dose unfractionated heparin (100 IU/kg/daily)

ELIGIBILITY:
Inclusion Criteria:

* Age between 4 and 60 years
* Short term non-tunneled percutaneous central venous catheter

Exclusion Criteria:

* Presence of a central venous catheter at admission
* Major blood coagulation disorders (platelet count < 50 x 10^9, disseminated intravascular coagulation)
* Absence of catheter-tip culture at the time of catheter removal

Ages: 4 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2005-05; Study Completion 2005-08

PRIMARY OUTCOMES:
Incidence of catheter-related bloodstream infection in 2 groups of patients with haemato-oncological disease
Group A: heparin impregnated catheters
Group B: continuous infusion of low dose unfractionated heparin (100IU/kg/d) through non-impregnated catheter.

SECONDARY OUTCOMES:
Analysis of variables that may be significant for the development of catheter-related bloodstream infection (catheter-related thrombosis; age; underlying disease; side of venous puncture; duration of catheterization)

CONTACTS AND LOCATIONS:
Overall Officials: Abderrahman Abdelkefi, MD, Principal Investigator — Centre National de Greffe de Moelle Osseuse
Locations (1):
- Centre National de Greffe de Moelle Osseuse, Tunis, Tunis Governorate, Tunisia